CLINICAL TRIAL: NCT01149525
Title: A Randomised, Double Blinded Cross-over Study Comparing the Efficacy of L-carnitine Versus Placebo in the Treatment of Fatigue in Multiple Sclerosis
Brief Title: Efficacy of L-carnitine Versus Placebo in the Treatment of Fatigue in Multiple Sclerosis
Acronym: FACTSEP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CHUBX 2009/13
Record Dates: First submitted 2010-06-21; First posted 2010-06-23 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis/complications; Fatigue Syndrome; Chronic/drug therapy
MeSH Terms: conditions — Multiple Sclerosis | interventions — Carnitine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): oral solution of L-Carnitine, 4g per day
  Interventions: Drug: L-Carnitine
- 2 (Placebo Comparator): Similar oral solution without L-Carnitine
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: L-Carnitine — 2g oral solution , twice per day (morning/evening), during 3 months
  Arms: 1
Drug: Placebo — oral solution, twice per day (morning/evening), during 3 months
  Arms: 2

SUMMARY:
The objective of this study is to evaluate the efficacy of L-carnitine versus placebo in the treatment of fatigue in multiple sclerosis patients. This study will randomize 60 patients in a cross-over design. This study is sponsored by academic French health institutions.

DETAILED DESCRIPTION:
Fatigue is one of the most frequent disabling symptom in Multiple Sclerosis (MS). L-Carnitine is currently used in the symptomatic treatment of fatigue after chemotherapy in patients with cancers. It is also empirically used by numerous MS centers in the treatment of fatigue. However, this practice is not evidence-based (Cochrane review 2010). This study will evaluate the efficacy of L-carnitine versus placebo in the treatment of fatigue in MS patients in a randomized double blind national multicenter cross-over trial.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and older
* Relapsing remitting (RR) secondary progressive (SP) or primary progressive multiple sclerosis according to McDonald 2005 (Polman) MS diagnostic criteria.
* Affected of fatigue for more than 3 months with global score on Modified Fatigue Impact Scale (MFIS)>45.
* Indication of treatment of fatigue to the appreciation of the neurologist.
* Expanded Disability Status Scale (EDSS) not exceeding 6.0.
* Information and comprehensive agreement signed by patient and the investigator.
* Subject affiliated to health insurance coverage.

Exclusion Criteria:

* Patients with serious unstable disease :

  * recurrent or serious relapses
  * rapidly ongoing disability impairment in the preceding 6 months
  * serious or non stabilized depression
* Patients starting a new disease modifying therapy, immunosuppression or antidepressant therapy less than 3 months ago or not stabilized.
* Patients with a treatment of fatigue or of other condition that may interfere with fatigue evaluation to the appreciation of the neurologist.
* Energy drinks consumption or toxicomania.
* All other reasons to the opinion of the neurologist that may impair study management, especially patient compliance, neuro-psychological disorders that may input questionnaires filling.
* Person under protection of the law.
* Participation in other clinical trials (allowing for exceptions, after recommendation from the scientific council).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2010-06; Primary Completion 2013-03 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Global score on the 21 item Modified Fatigue Impact Scale (MFIS, translated and validated in French). | Three months and nine months (2 periods of 3 months on treatment/placebo separated by a wash-out period of 3 months)

SECONDARY OUTCOMES:
Fatigue Severity Scale (FSS) | Three and nine months
Fatigue Visual Analogic Scale (VAS) | Three and nine months
physical dimension scale of MFIS | Three and nine months
SEP59 scale of quality of life (Multiple Sclerosis Quality Of Life scale validated in french) | Three and nine months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe OUALLET, MD-PhD, Principal Investigator — University Hospital Bordeaux, France; Geneviève CHENE, MD-PhD, Study Chair — USMR (University Hospital, Bordeaux)
Locations (6):
- France (6):
  - University Hospital, Hospital Pellegrin, Bordeaux
  - University Hospital, Fort de France
  - University Hospital, Hospital Dupuytren, Limoges
  - University Hospital, Hospital Central, Nancy
  - University Hospital, Hospital Laënnec, Nantes
  - University Hospital, Hospital Pasteur, Nice

REFERENCES:
- [Background] Tejani AM, Wasdell M, Spiwak R, Rowell G, Nathwani S. Carnitine for fatigue in multiple sclerosis. Cochrane Database Syst Rev. 2010 Feb 17;(2):CD007280. doi: 10.1002/14651858.CD007280.pub2. PMID 20166093
- [Background] Bakshi R. Fatigue associated with multiple sclerosis: diagnosis, impact and management. Mult Scler. 2003 Jun;9(3):219-27. doi: 10.1191/1352458503ms904oa. PMID 12814166
- [Background] Filippi M, Rocca MA, Colombo B, Falini A, Codella M, Scotti G, Comi G. Functional magnetic resonance imaging correlates of fatigue in multiple sclerosis. Neuroimage. 2002 Mar;15(3):559-67. doi: 10.1006/nimg.2001.1011. PMID 11848698
- [Background] Oken BS, Kishiyama S, Zajdel D, Bourdette D, Carlsen J, Haas M, Hugos C, Kraemer DF, Lawrence J, Mass M. Randomized controlled trial of yoga and exercise in multiple sclerosis. Neurology. 2004 Jun 8;62(11):2058-64. doi: 10.1212/01.wnl.0000129534.88602.5c. PMID 15184614
- [Background] Pucci E, Branas P, D'Amico R, Giuliani G, Solari A, Taus C. Amantadine for fatigue in multiple sclerosis. Cochrane Database Syst Rev. 2007 Jan 24;2007(1):CD002818. doi: 10.1002/14651858.CD002818.pub2. PMID 17253480
- [Background] Krupp LB, Coyle PK, Doscher C, Miller A, Cross AH, Jandorf L, Halper J, Johnson B, Morgante L, Grimson R. Fatigue therapy in multiple sclerosis: results of a double-blind, randomized, parallel trial of amantadine, pemoline, and placebo. Neurology. 1995 Nov;45(11):1956-61. doi: 10.1212/wnl.45.11.1956. PMID 7501140
- [Background] van Diemen HA, Polman CH, van Dongen TM, van Loenen AC, Nauta JJ, Taphoorn MJ, van Walbeek HK, Koetsier JC. The effect of 4-aminopyridine on clinical signs in multiple sclerosis: a randomized, placebo-controlled, double-blind, cross-over study. Ann Neurol. 1992 Aug;32(2):123-30. doi: 10.1002/ana.410320203. PMID 1510353
- [Background] Stankoff B, Waubant E, Confavreux C, Edan G, Debouverie M, Rumbach L, Moreau T, Pelletier J, Lubetzki C, Clanet M; French Modafinil Study Group. Modafinil for fatigue in MS: a randomized placebo-controlled double-blind study. Neurology. 2005 Apr 12;64(7):1139-43. doi: 10.1212/01.WNL.0000158272.27070.6A. PMID 15824337
- [Background] Tomassini V, Pozzilli C, Onesti E, Pasqualetti P, Marinelli F, Pisani A, Fieschi C. Comparison of the effects of acetyl L-carnitine and amantadine for the treatment of fatigue in multiple sclerosis: results of a pilot, randomised, double-blind, crossover trial. J Neurol Sci. 2004 Mar 15;218(1-2):103-8. doi: 10.1016/j.jns.2003.11.005. PMID 14759641
- [Background] Wingerchuk DM, Benarroch EE, O'Brien PC, Keegan BM, Lucchinetti CF, Noseworthy JH, Weinshenker BG, Rodriguez M. A randomized controlled crossover trial of aspirin for fatigue in multiple sclerosis. Neurology. 2005 Apr 12;64(7):1267-9. doi: 10.1212/01.WNL.0000156803.23698.9A. PMID 15824361
- [Background] Lebrun C, Alchaar H, Candito M, Bourg V, Chatel M. Levocarnitine administration in multiple sclerosis patients with immunosuppressive therapy-induced fatigue. Mult Scler. 2006 Jun;12(3):321-4. doi: 10.1191/135248506ms1275oa. PMID 16764345
- [Background] Pittion-Vouyovitch S, Debouverie M, Guillemin F, Vandenberghe N, Anxionnat R, Vespignani H. Fatigue in multiple sclerosis is related to disability, depression and quality of life. J Neurol Sci. 2006 Apr 15;243(1-2):39-45. doi: 10.1016/j.jns.2005.11.025. Epub 2006 Jan 24. PMID 16434057
- [Background] Debouverie M, Pittion S. [Fatigue and episodic exhaustion as a feature of multiple sclerosis]. Rev Neurol (Paris). 2006 Mar;162(3):295-7. doi: 10.1016/s0035-3787(06)75015-9. No abstract available. French. PMID 16585884
- [Background] Richardson BA, Flack VF. The analysis of incomplete data in the three-period two-treatment cross-over design for clinical trials. Stat Med. 1996 Jan 30;15(2):127-43. doi: 10.1002/(SICI)1097-0258(19960130)15:23.0.CO;2-D. PMID 8614750
- [Background] GRIZZLE JE. THE TWO-PERIOD CHANGE-OVER DESIGN AN ITS USE IN CLINICAL TRIALS. Biometrics. 1965 Jun;21:467-80. No abstract available. PMID 14338679
- [Background] Kieser M, Friede T. Re-calculating the sample size in internal pilot study designs with control of the type I error rate. Stat Med. 2000 Apr 15;19(7):901-11. doi: 10.1002/(sici)1097-0258(20000415)19:73.0.co;2-l. PMID 10750058
- [Background] Graziano F, Bisonni R, Catalano V, Silva R, Rovidati S, Mencarini E, Ferraro B, Canestrari F, Baldelli AM, De Gaetano A, Giordani P, Testa E, Lai V. Potential role of levocarnitine supplementation for the treatment of chemotherapy-induced fatigue in non-anaemic cancer patients. Br J Cancer. 2002 Jun 17;86(12):1854-7. doi: 10.1038/sj.bjc.6600413. PMID 12085175
- [Background] Plioplys AV, Plioplys S. Amantadine and L-carnitine treatment of Chronic Fatigue Syndrome. Neuropsychobiology. 1997;35(1):16-23. doi: 10.1159/000119325. PMID 9018019
- [Background] Debouverie M, Pittion-Vouyovitch S, Louis S, Guillemin F. Validity of a French version of the fatigue impact scale in multiple sclerosis. Mult Scler. 2007 Sep;13(8):1026-32. doi: 10.1177/1352458507077942. PMID 17895294
- [Background] Montel SR, Bungener C. Coping and quality of life in one hundred and thirty five subjects with multiple sclerosis. Mult Scler. 2007 Apr;13(3):393-401. doi: 10.1177/1352458506071170. Epub 2007 Jan 29. PMID 17439909
- [Background] Cruciani RA, Dvorkin E, Homel P, Malamud S, Culliney B, Lapin J, Portenoy RK, Esteban-Cruciani N. Safety, tolerability and symptom outcomes associated with L-carnitine supplementation in patients with cancer, fatigue, and carnitine deficiency: a phase I/II study. J Pain Symptom Manage. 2006 Dec;32(6):551-9. doi: 10.1016/j.jpainsymman.2006.09.001. PMID 17157757
- [Background] Gramignano G, Lusso MR, Madeddu C, Massa E, Serpe R, Deiana L, Lamonica G, Dessi M, Spiga C, Astara G, Maccio A, Mantovani G. Efficacy of l-carnitine administration on fatigue, nutritional status, oxidative stress, and related quality of life in 12 advanced cancer patients undergoing anticancer therapy. Nutrition. 2006 Feb;22(2):136-45. doi: 10.1016/j.nut.2005.06.003. PMID 16459226
- [Background] Neri S, Pistone G, Saraceno B, Pennisi G, Luca S, Malaguarnera M. L-carnitine decreases severity and type of fatigue induced by interferon-alpha in the treatment of patients with hepatitis C. Neuropsychobiology. 2003;47(2):94-7. doi: 10.1159/000070016. PMID 12707492
- [Background] Rebouche CJ. Kinetics, pharmacokinetics, and regulation of L-carnitine and acetyl-L-carnitine metabolism. Ann N Y Acad Sci. 2004 Nov;1033:30-41. doi: 10.1196/annals.1320.003. PMID 15591001
- [Background] Plioplys AV, Plioplys S. Serum levels of carnitine in chronic fatigue syndrome: clinical correlates. Neuropsychobiology. 1995;32(3):132-8. doi: 10.1159/000119226. PMID 8544970
- [Background] Cruciani RA, Dvorkin E, Homel P, Culliney B, Malamud S, Shaiova L, Fleishman S, Lapin J, Klein E, Lesage P, Portenoy R, Esteban-Cruciani N. L-carnitine supplementation for the treatment of fatigue and depressed mood in cancer patients with carnitine deficiency: a preliminary analysis. Ann N Y Acad Sci. 2004 Nov;1033:168-76. doi: 10.1196/annals.1320.016. PMID 15591014
- [Background] Taglialatela G, Navarra D, Cruciani R, Ramacci MT, Alema GS, Angelucci L. Acetyl-L-carnitine treatment increases nerve growth factor levels and choline acetyltransferase activity in the central nervous system of aged rats. Exp Gerontol. 1994 Jan-Feb;29(1):55-66. doi: 10.1016/0531-5565(94)90062-0. PMID 8187841